CLINICAL TRIAL: NCT05126004
Title: Azacitidine (AZA) Combined With N-Acetyl-L-cysteine (NAC) for Prolonged Isolated Thrombocytopenia (PIT) After Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: AZA Combined With NAC for PIT After HSCT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOOCHOW-HY-2021-2
Record Dates: First submitted 2021-07-30; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-04

CONDITIONS: Thrombocytopenia, Isolated; Stem Cell Transplant Complications
Keywords: Azacitidine; N-Acetyl-L-cysteine; Prolonged Isolated Thrombocytopenia; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Thrombocytopenia | interventions — Azacitidine; Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Arm1: Control Arm2:AZA+NAC
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): receive supportive care
- AZA+NAC group (Experimental): AZA 50mg Subcutaneous daily d1-d5 + NAC 600mg oral bid d1-28， 28 days for one cycle
  Interventions: Drug: Azacitidine; Drug: N Acetyl L Cysteine

INTERVENTIONS:
Drug: Azacitidine — 28 days for one cycle, evaluation post 3 cycles of treatment. Continue if response exists, otherwise, quit the trial and seek for other therapies.
  Other Names: AZA
  Arms: AZA+NAC group
Drug: N Acetyl L Cysteine — 28 days for one cycle, evaluation post 3 cycles of treatment. Continue if response exists, otherwise, quit the trial and seek for other therapies.
  Other Names: NAC
  Arms: AZA+NAC group

SUMMARY:
Prolonged isolated thrombocytopenia (PIT) that is refractory to conventional treatments has remained a critical complication after allogeneic hematopoietic cell transplantation since decades years ago. Recombinant human thrombopoietin (rhTPO) is the main therapy in clinical practice, but remains low efficiency for PIT. Demethylating drugs have shown thier potential in high-risk myelodysplastic syndromes (MDS) and acte myeloid leukemia (AML). In addition, decitabine has demonstrated its efficacy of over 70% for response rate in treatment for PIT in early clinical trials with elusive mechanism. Preliminary experiments revealed that PIT was associated with abnormality of oxidation microenvironment, and N-Acetyl-L-cysteine (NAC) was the most commonly used antioxidant. Therefore, the investigators have been wondering whether Azacitidine in combination with NAC could improve PIT post HSCT and explore the possible mechanism of it.

DETAILED DESCRIPTION:
Prolonged isolated thrombocytopenia (PIT) that is refractory to conventional treatments has remained a critical complication after allogeneic hematopoietic cell transplantation since decades years ago. Recombinant human thrombopoietin (rhTPO) is the main therapy in clinical practice, but remains low efficiency for PIT. Demethylating drugs have shown thier potential in high-risk myelodysplastic syndromes (MDS) and acte myeloid leukemia (AML). In addition, decitabine has demonstrated its efficacy of over 70% for response rate in treatment for PIT in early clinical trials with elusive mechanism. Preliminary experiments revealed that PIT was associated with abnormality of oxidation microenvironment, and N-Acetyl-L-cysteine (NAC) was the most commonly used antioxidant. Furthermore, AZA had shown its potential in immune regulation. Therefore, the investigators have been wondering whether Azacitidine in combination with NAC could improve PIT post HSCT and explore the possible mechanism of it.

ELIGIBILITY:
Inclusion Criteria:

* Platelet count ≤ 30 × 10^9/L persistently at day 60 post-HSCT or later;
* Neutrophil and hemoglobin were well recovered;
* Full donor chimerism was achieved;

Exclusion Criteria:

* Patients with malignancy relapse;
* Active infections;
* Grade Ⅲ-Ⅳ acute graft-versus-host disease or severe chronic graft-versus-host disease according to National Institute of Health criteria;
* Severe organ damage;
* Thrombosis requiring treatment;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
platelet reconstruction | From date of randomization until the date of platelet reconstruction, assessed up to 100 days
  platelet count above 50*10^9/L independent of transfusion

SECONDARY OUTCOMES:
overall survival | From date of randomization until the date of death from any cause, assessed up to 1 year
  the time from the date of day 1 post HSCT to the date of death due to any cause
overall response rate | From date of randomization until the date of platelet count between 30*10^9/L and 50*10^9/L, assessed up to 100 days
  platelet count evaluating above 30*10^9/L but below 50*10^9/L independent of platelet transfusion

OTHER OUTCOMES:
infection | From date of randomization until the date of diagnose of infection, assessed up to 100 days
  clinical diagnose of infection or evidence of next generation of sequencing（NGS）of body fluid or CT or culture of samples collected from patients
Severe adverse events | From date of randomization until the date of occurrence of any severe adverse event, assessed up to 100 days
  any events that prevent the clinical trial continue besides hepatic injury renal function impairment, et al.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] First LR, Smith BR, Lipton J, Nathan DG, Parkman R, Rappeport JM. Isolated thrombocytopenia after allogeneic bone marrow transplantation: existence of transient and chronic thrombocytopenic syndromes. Blood. 1985 Feb;65(2):368-74. PMID 3881142
- [Background] Bruno B, Gooley T, Sullivan KM, Davis C, Bensinger WI, Storb R, Nash RA. Secondary failure of platelet recovery after hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2001;7(3):154-62. doi: 10.1053/bbmt.2001.v7.pm11302549.
- [Background] Wang H, Huang M, Zhao Y, Qi JQ, Chen C, Tang YQ, Qiu HY, Fu CC, Tang XW, Wu DP, Ruan CG, Han Y. Recombinant Human Thrombopoietin Promotes Platelet Engraftment and Improves Prognosis of Patients with Myelodysplastic Syndromes and Aplastic Anemia after Allogeneic Hematopoietic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2017 Oct;23(10):1678-1684. doi: 10.1016/j.bbmt.2017.06.010. Epub 2017 Jun 19. PMID 28642072
- [Background] Zhao X, Zhao X, Huo M, Fan Q, Pei X, Wang Y, Zhang X, Xu L, Huang X, Liu K, Chang Y. Donor-Specific Anti-Human Leukocyte Antigen Antibodies Predict Prolonged Isolated Thrombocytopenia and Inferior Outcomes of Haploidentical Hematopoietic Stem Cell Transplantation. J Immunol Res. 2017;2017:1043836. doi: 10.1155/2017/1043836. Epub 2017 Apr 16. PMID 28484721
- [Background] Ramirez P, Brunstein CG, Miller B, Defor T, Weisdorf D. Delayed platelet recovery after allogeneic transplantation: a predictor of increased treatment-related mortality and poorer survival. Bone Marrow Transplant. 2011 Jul;46(7):981-6. doi: 10.1038/bmt.2010.218. Epub 2010 Oct 4. PMID 20921943
- [Background] Tang Y, Chen J, Liu Q, Chu T, Pan T, Liang J, He XF, Chen F, Yang T, Ma X, Wu X, Hu S, Cao X, Hu X, Hu J, Liu Y, Qi J, Shen Y, Ruan C, Han Y, Wu D. Low-dose decitabine for refractory prolonged isolated thrombocytopenia after HCT: a randomized multicenter trial. Blood Adv. 2021 Mar 9;5(5):1250-1258. doi: 10.1182/bloodadvances.2020002790. PMID 33646303
- [Background] Mohyeldin A, Garzon-Muvdi T, Quinones-Hinojosa A. Oxygen in stem cell biology: a critical component of the stem cell niche. Cell Stem Cell. 2010 Aug 6;7(2):150-61. doi: 10.1016/j.stem.2010.07.007. PMID 20682444
- [Background] Chen S, Su Y, Wang J. ROS-mediated platelet generation: a microenvironment-dependent manner for megakaryocyte proliferation, differentiation, and maturation. Cell Death Dis. 2013 Jul 11;4(7):e722. doi: 10.1038/cddis.2013.253. PMID 23846224
- [Background] Kong Y, Shi MM, Zhang YY, Cao XN, Wang Y, Zhang XH, Xu LP, Huang XJ. N-acetyl-L-cysteine improves bone marrow endothelial progenitor cells in prolonged isolated thrombocytopenia patients post allogeneic hematopoietic stem cell transplantation. Am J Hematol. 2018 Jul;93(7):931-942. doi: 10.1002/ajh.25056. Epub 2018 Feb 24. PMID 29396859
- [Background] Han Y, Tang Y, Chen J, Liang J, Ye C, Ruan C, Wu D. Low-Dose Decitabine for Patients With Thrombocytopenia Following Allogeneic Hematopoietic Stem Cell Transplantation: A Pilot Therapeutic Study. JAMA Oncol. 2015 May;1(2):249-51. doi: 10.1001/jamaoncol.2014.316. No abstract available. PMID 26181032
- [Background] Zhou H, Hou Y, Liu X, Qiu J, Feng Q, Wang Y, Zhang X, Min Y, Shao L, Liu X, Li G, Li L, Yang L, Xu S, Ni H, Peng J, Hou M. Low-dose decitabine promotes megakaryocyte maturation and platelet production in healthy controls and immune thrombocytopenia. Thromb Haemost. 2015 May;113(5):1021-34. doi: 10.1160/TH14-04-0342. Epub 2015 Jan 8. PMID 25566808

DOCUMENTS (1):
  • Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT05126004/ICF_000.pdf